CLINICAL TRIAL: NCT03247387
Title: Evaluation of the eON-OFF Mobile Application and Four Actigraphy Devices in Subjects With Parkinson's Disease
Brief Title: eOnOff - D1 Extension
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Kevin C.Thomas, Assistant Professor, Anatomy & Neurobiology, Boston University
Other Study IDs: H-35364
Record Dates: First submitted 2017-08-07; First posted 2017-08-11 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
Keywords: Wearable device; Patient monitor
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MC10 BioStampRC — Subjects will fill out electronic diaries on a provisioned iPhone to capture "On" versus "Off" time on a daily basis while at home. In addition, subjects will be asked to wear three actigraphy devices.
Device: APDM actigraphy device — Subjects will fill out electronic diaries on a provisioned iPhone to capture "On" versus "Off" time on a daily basis while at home. In addition, subjects will be asked to wear three actigraphy devices.
Device: GENEActiv watch — Subjects will fill out electronic diaries on a provisioned iPhone to capture "On" versus "Off" time on a daily basis while at home. In addition, subjects will be asked to wear three actigraphy devices.

SUMMARY:
Clinical assessments can only offer a snapshot of daily life with Parkinson's Disease, while wearable devices can offer immensely more information that can improve the understanding of this disease. With recent advancements in technology, investigators are now able to use watch-like devices to more effectively measure the symptoms of Parkinson's Disease outside of the doctor's office. The present study is designed to evaluate the usability, applicability, and interpretability of an electronic VA Patient Motor Diary (eON-OFF), MC10 BioStampRC actigraphy sensor, APDM actigraphy sensor and the GENEActiv Watch in persons with Parkinson's Disease. There is no placebo/control group.

DETAILED DESCRIPTION:
The proposed study will be comprised of at least four sessions in the Spivack Center (Rm. X-140) on separate days (not counting recruitment, screening, or consent activities), each lasting approximately 1-2 hours. Subjects will commence a 1-week testing period during which they will wear the 3 actigraphy devices in their normal schedule and daily environment. On Days 2, 3, 4, and 5, subjects will use the eON-OFF motor diary application to select their current Parkinson state (e.g. "on", "off"). ON and OFF states are subjective measures identified by subjects, and are commonly used words in Parkinson's Disease treatment and research to describe symptom states. Symptom severity is directly linked to medication effectiveness. "On" is when the medication is working and symptoms are not severe or troublesome. "Off" is when medication has worn off, and symptom severity increases. Subjects will also use the eON-OFF motor diary application to verbally record symptomology every 30 minutes while awake. Subjects will complete paper VA Patient Motor Diaries to record ON and OFF states on Day 2, Day 3, and Day 4. Subjects will then complete the outlined set of activities during Phase I in a second phase to take place approximately one month later. All questionnaires, training and interviews will be administered one-on-one by a trained research assistant. All UPDRS' will be administered by a clinician. Ideally, subjects will be administered the study activities on the days listed above, but they are allowed a flexibility of +/- 4 days for scheduling appointments.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported clinical diagnosis of Parkinson's disease consistent with the United Kingdom (UK) Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria.
* Self-reported ability to recognize their "wearing off" symptoms and confirmation that they usually improve after their next dose of Parkinson's disease medication.
* Parkinson's disease Hoehn & Yahr Stage less than or equal to III (assessed while the patient is "ON").
* Currently responding to L-Dopa therapy. On a stable dose of L-Dopa (or L-Dopa equivalent) of at least 300 mg total daily dose for at least 28 days prior to Day 1, in conjunction with a dopa decarboxylase inhibitor (e.g., L-Dopa/carbidopa or L-Dopa/benserazide) divided in at least 3 divided doses per day.
* 45-75 years old
* Able to understand and cooperate with study procedures and give informed consent.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* Body Mass Index (BMI) of 17.5 to 35 kg/m2; and a total body weight of greater than or equal to 45kg.
* Native English speaker or demonstrated fluency in English.
* Normal or corrected-to-normal vision
* A score of greater than or equal to 26 on the Mini Mental State Examination (MMSE).
* A score of 49 on the Green Form of the WRAT-4 Word Reading Subtest (equivalent to 8th grade reading level)

Exclusion Criteria:

* Treatment with an investigational drug within 30 days of Day 1 of study activities.
* Diagnosis of moderate to severe alcohol use disorder within 6 months of the screening as disclosed by the subject
* Employees, student, or advisee of the Principal Investigator
* History of head injury with clinically significant sequelae (e.g. loss of consciousness for greater than 15 minutes).
* DSM-V diagnosis of current, or history of, neurological disease (except for Parkinson's disease), Schizophrenia Spectrum or Other Psychotic disorders, or Bipolar and Related Disorders as disclosed by the subject.
* Subjects with cardiac pacemakers, electronic pumps, or any other implanted medical devices, including deep brain stimulation devices.
* Women of childbearing age will be required to undergo a pregnancy test to rule out a possible pregnancy.
* Allergy to adhesives or silicone

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with Parkinson's disease.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Assessment of eON-OFF mobile application ("eON-OFF app") in PD subjects. | 2 week long periods spaced a month apart
  Subjects will use the eON-OFF motor diary application to select their current Parkinson state (e.g. "on", "off"). Subjects will also use the eON-OFF motor diary application to verbally record symptomology every 30 minutes while awake.

SECONDARY OUTCOMES:
Equivalence testing of the eON-OFF app on provisioned devices against established paper-based clinical assessment. | 2 week long periods spaced a month apart
  Subjects will complete paper VA Patient Motor Diaries to record ON and OFF states. ON and OFF states are subjective measures identified by subjects, and are commonly used words in Parkinson's Disease treatment and research to describe symptom states.
Evaluation of the usability and applicability of 3 wearable sensor systems in assessing clinical measures of PD. | 2 week long periods spaced a month apart
  Subjects will undergo two, 1-week testing periods during which they will wear the 3 actigraphy devices in their normal schedule and daily environment.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Thomas, PhD MBA, Principal Investigator — BU Anatomy and Neurology Dept, Evans Biomedical Research Center
Locations (1):
- Evans Biomedical Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No